CLINICAL TRIAL: NCT07058506
Title: Evaluation of Non-invasive Control Interfaces for Operating Assistive Devices for Tetraplegic Individuals
Brief Title: Control Interfaces for Operating Assistive Devices
Acronym: SENSORS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Bouffard Vercelli - USSAP (Other)
Collaborators: NEURINNOV (Unknown); Institut National de Recherche en Informatique et en Automatique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-A01014-43; 101099916 (Other Grant/Funding Number: HORIZON-EIC-2022-PATHFINDEROPEN-01)
Record Dates: First submitted 2025-06-06; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Tetraplegia
Keywords: Tetraplegia; Non-invasive control interfaces; Sensors
MeSH Terms: conditions — Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with complete tetraplegia AIS A or B, with a neurological level ≥ C7 (Experimental)
  Interventions: Device: Comparison of 5 interfaces used to capture user intent to operate a neuroprosthesis

INTERVENTIONS:
Device: Comparison of 5 interfaces used to capture user intent to operate a neuroprosthesis — No intervention

SUMMARY:
Neurinnov, in collaboration with the CBV USSAP center and the CAMIN INRIA team, has conducted clinical investigations using various control interfaces, including EMG, IMU, contact sensors, and voice commands, to operate a motor neuroprosthesis. This neuroprosthesis is based on neural electrical stimulation, enabling the activation of multiples muscles via a single electrode. The clinical investigations have successfully demonstrated the feasibility of achieving grasping movements induced by neural electrical stimulation, which are controlled by the participant through external interfaces.

These external interfaces were based on existing technologies but were only suitable for research purposes due to their lack of portability. The current investigation aims to validate fully portable interfaces designed by Neurinnov, which are intended to be integral components of a future medical device that includes an implanted stimulator and its neural electrodes. The study's goal is to demonstrate that these interfaces can be used by participants with sufficient success rate (clinical performance) to support daily use.

Our main hypothesis is that the participants can effectively use at least two of the six control interfaces presented to them to detect their intention to perform a motor action within a software environment under constant conditions. These interfaces include voice commands, inertial measurement unit (IMU) sensors, surface electromyography (EMG) sensors, switch, joystick, and earswitch.

DETAILED DESCRIPTION:
Various control interfaces (CIs) are used to capture user intent for operating assistive devices. In recent years, several methods have been developed to detect user intent for controlling invasive motor neuroprostheses for upper limbs. The Freehand System® utilized an external shoulder position sensor on the contralateral side to detect user intent and control hand grasp stimulation. In some studies, a switch was integrated with the sensor to turn the system on and off and to select the type of grasp (palmar or lateral). Brain-computer interface (BCI) systems based on electroencephalography (EEG) have also been employed. The Implantable Stimulator-Telemeter ('IST-10'), the second generation of the Freehand, had ten stimulation channels and was used with an implantable joint angle sensor. The third generation, the Implanted Stimulator Telemeter (IST-12), used myoelectric signals. However, no direct comparison has been made between these different modalities, nor has their relevance been determined.

Therefore, this study aims to evaluate the performance (efficacy: reliability and precision) of six non-invasive control interfaces. The efficacy criterion is defined by the ability to reliably and accurately control a motor action as illustrated by software on a screen. The six control interfaces are: (1) inertial measurement unit (IMU) sensors that record movements of the contralateral shoulder; (2) surface electromyography (EMG) sensors that capture voluntary muscle contractions of the contralateral limb; (3) a pressure sensor button (switch sensor); (4) a pressure sensor joystick (joystick sensor); (5) a voice recognition sensor (voice sensor) that incorporates a machine learning model capable of recognizing specific words spoken by the participant; and (6) an Ear-Switch® sensor that detects movements of a muscle inside the ear, the tensor tympani.

The study will be conducted over six sessions:

* (V1) Selection Visit: The selection visit will be conducted by the coordinating investigator, who will monitor the participant throughout the trial.
* (V2) Inclusion Visit: This visit will include:

  * Clinical examination
  * Collection of the signed consent form
  * Audio recordings of key words to personalize the speech recognition algorithms
* (V3 to V5) Experimental Visits:

  * V3: Evaluation of all six control interfaces.
  * V4: Detailed assessment of the two best-mastered control interfaces, both separately and in combination (bimodal use).
  * V5: Intensity modulation visit, assessing the participant's ability to reliably and accurately reach target static and dynamic intensity levels (as shown on a screen) using two of the interfaces.
* (V6) End-of-Study Visit: This final visit will consist of a clinical and psychological follow-up consultation to ensure the absence of any adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury defined by an AIS A, B or C score (AIS A, B or C): complete or incomplete motor deficit below the lesion. This is a standard for describing spinal cord injuries that has been internationally agreed upon.
* Spinal cord injury at the neurological level > C7
* Age greater than or equal to 18 and less than or equal to 80 years
* A history of more than 3 months of neurological stability, with no changes in muscle testing.
* Participants capable of following instructions for testing and providing feedback on the use of the device.
* Participants who have signed the informed consent form to participate in the study after being fully informed.
* Participants affiliated with a social security system (either as a beneficiary or a dependent), excluding those covered by State Medical Aid (AME).

Exclusion Criteria:

* Participant deprived of liberty (by judicial or administrative decision).
* Adult participants are under legal protection or unable to provide informed consent.
* Participation in another ongoing clinical trial.
* Unstable psychiatric condition.
* Severe cognitive impairment.
* Unstable acute medical condition
* Insufficient proficiency in spoken and written French.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy indicators | At Day 1
  Success rate: describes the ability of a control interface to execute requested functions under specified conditions Evaluation criterion: (Number of correctly recognized commands) / (Number of correctly recognized commands + Number of incorrectly recognized commands). Rate in percentage %

SECONDARY OUTCOMES:
Time workload indicators | At Day 1
  Latency between the user's actual intention and its detection, measured in seconds.
Indicator of feasibility: Ease of installation, calibration, and learning of each control interface (CI) | At Day 2 for the points 1, 2 and 3 and at Day 3 for the point 4
  Evaluation criterion: Time tracked by the sensor control software, measured in minutes.
Indicator of feasibility: Ease of placing the control interface | At Day 2 for the points 1, 2 and 3 and at Day 3 for the point 4
  Evaluation criterion: The number of times a third party (participant's caregiver or clinician) needed physical assistance and/or requested additional instructions to position the sensor.
Indicator of feasibility: Ease of learning to use the control interface | At Day 2 for the points 1, 2 and 3 and at Day 3 for the point 4
  Evaluation criterion: The number of repetitions required for the participant to learn the interface.
  At Day 2 for the points 1, 2 and 3 and at Day 3 for the point 4
Indicator of feasibility: User feedback concerning usability of the control interface | At Day 2 for the points 1, 2 and 3 and at Day 3 for the point 4
  Evaluation criterion: System Usability Scale French Version (F-SUS) Score min: 10 and score max: 50
Indicator of tolerance : Pain experienced during and after using the interface | During the experimentation at Day 2 and 3
  Evaluation criterion: visual analog scale (VAS) ranging from 0 to 10.
Indicator of tolerance : Adverse effects | During the experimentation at Day 2 and 3
  Adverse effects encountered during and after using the interface.
Indicators of satisfaction, comfort, pleasure of use and subjective workload | At Day 3
  User satisfaction with the control interface (CI) Evaluation criterion: Quebec User Evaluation of Satisfaction with Assistive Technology (French version = ESAT) . Score min : 12 and score max: 60
Indicators of satisfaction, comfort, pleasure of use and subjective workload | At Day 3
  Enjoyability of the control interface, reflecting the user's mood, motivation, or frustration.
  Evaluation criterion: appropriate section of the questionnaire National Aeronautics and Space Administration Task Load Index (NASA-TLX). For each item, the score min is 0 and max 100
Indicators of satisfaction, comfort, pleasure of use and subjective workload | At Day 3
  User perception of subjective workload Evaluation criterion: questionnaire National Aeronautics and Space Administration Task Load Index (NASA-TLX). For each item, the score min is 0 and max 100
Indicators that a static and dynamic intensity value has been reached in a predetermined time (difference between target and initial value) | At Day 7
  Static trial: successful target acquisition within the allotted time (acquisition time in seconds).
Indicators that a static and dynamic intensity value has been reached in a predetermined time (difference between target and initial value) | At Day 7
  2. Dynamic trial: the user-controlled value remains within a 10% margin of error relative to the reference value throughout the trial. (margin of error in percentage %)

CONTACTS AND LOCATIONS:
Overall Officials: Charles FATTAL, MD, PhD, Principal Investigator — Centre Bouffard Vercelli - USSAP
Locations (1):
- Rehabilitation Center Bouffard-Vercelli USSAP, Perpignan, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fattal C, Teissier J, Geffrier A, Fonseca L, William L, Andreu D, Guiraud D, Azevedo-Coste C. Restoring Hand Functions in People with Tetraplegia through Multi-Contact, Fascicular, and Auto-Pilot Stimulation: A Proof-of-Concept Demonstration. J Neurotrauma. 2022 May;39(9-10):627-638. doi: 10.1089/neu.2021.0381. Epub 2022 Feb 2. PMID 35029125
- [Background] Fonseca L, Guiraud D, Hiairrassary A, Fattal C, Azevedo-Coste C. A Residual Movement Classification Based User Interface for Control of Assistive Devices by Persons With Complete Tetraplegia. IEEE Trans Neural Syst Rehabil Eng. 2022;30:569-578. doi: 10.1109/TNSRE.2022.3156269. Epub 2022 Mar 21. PMID 35235517
- [Background] Tigra W, Dali M, William L, Fattal C, Gelis A, Divoux JL, Coulet B, Teissier J, Guiraud D, Azevedo Coste C. Selective neural electrical stimulation restores hand and forearm movements in individuals with complete tetraplegia. J Neuroeng Rehabil. 2020 May 19;17(1):66. doi: 10.1186/s12984-020-00676-4. PMID 32429963
- [Background] Fonseca L, Bo A, Guiraud D, Navarro B, Gelis A, Azevedo-Coste C. Investigating Upper Limb Movement Classification on Users with Tetraplegia as a Possible Neuroprosthesis Interface. Annu Int Conf IEEE Eng Med Biol Soc. 2018 Jul;2018:5053-5056. doi: 10.1109/EMBC.2018.8513418. PMID 30441476
- [Background] Fonseca L, Tigra W, Navarro B, Guiraud D, Fattal C, Bo A, Fachin-Martins E, Leynaert V, Gelis A, Azevedo-Coste C. Assisted Grasping in Individuals with Tetraplegia: Improving Control through Residual Muscle Contraction and Movement. Sensors (Basel). 2019 Oct 18;19(20):4532. doi: 10.3390/s19204532. PMID 31635286
- [Background] Coste CA, William L, Fonseca L, Hiairrassary A, Andreu D, Geffrier A, Teissier J, Fattal C, Guiraud D. Activating effective functional hand movements in individuals with complete tetraplegia through neural stimulation. Sci Rep. 2022 Oct 6;12(1):16189. doi: 10.1038/s41598-022-19906-x. PMID 36202865